CLINICAL TRIAL: NCT02937428
Title: To Look or Not to Look? Pilot Study of the Effectiveness of a Simple Psychological Intervention in Reducing Vaccination Pain and Fear in Adult
Brief Title: To Look or Not to Look at the Needle During Vaccination
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Anna Taddio, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33392
Record Dates: First submitted 2016-10-13; First posted 2016-10-18 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Vaccination
Keywords: vaccination; pain; fear; psychological intervention
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Look away and prefer to look (Experimental): Participant who is self-identified as preferring to look at the needle is randomized to look away from the needle during vaccination
  Interventions: Behavioral: Look away from the needle
- Look at needle and prefer to look (Active Comparator): Participant who is self-identified as preferring to look at the needle is randomized to look at the needle during vaccination
  Interventions: Behavioral: Look at the needle
- Look away and prefer to look away (Experimental): Participant who is self-identified as preferring to look away from the needle is randomized to look away from the needle during vaccination
  Interventions: Behavioral: Look away from the needle
- Look at needle and prefer to look away (Active Comparator): Participant who is self-identified as preferring to look away from the needle is randomized to look at the needle during vaccination
  Interventions: Behavioral: Look at the needle

INTERVENTIONS:
Behavioral: Look away from the needle — Participant looks away from the needle during vaccination
  Arms: Look away and prefer to look; Look away and prefer to look away
Behavioral: Look at the needle — Participant looks at the needle during vaccination
  Arms: Look at needle and prefer to look; Look at needle and prefer to look away

SUMMARY:
It is common for people to advise individuals undergoing vaccination to look away from the needle to make them hurt less and be less scary. However, this advice is not backed up by research evidence. the purpose of this study is to learn about how looking away vs. looking at the needle during vaccination makes people feel. People will be randomized to 1 of 2 groups: look at the needle, look away. Then they will undergo vaccination and report on pain and fear experienced.

DETAILED DESCRIPTION:
It is common for people to advise individuals undergoing vaccination to look away from the needle to make them hurt less and be less scary. However, this advice is not backed up by experimental research evidence. It is possible that looking away acts as a distraction and takes attention away from the needle, thus reducing pain. However, it is also possible that looking at the needle is better because it prevents people's imaginations from making them think it is worse than it actually is. To our knowledge, this is the first first randomized study to examine the effect of looking away vs. looking at the needle on pain and fear experienced during vaccinations. Adult university students undergoing routine flu vaccination will be included.

ELIGIBILITY:
Inclusion Criteria:

* undergraduate and graduate students at the University of Toronto's Leslie Dan Faculty of Pharmacy undergoing flu vaccination

Exclusion Criteria:

* less than 18 years of age or prior participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Pain | immediately after vaccination (<5 minutes)
  self-reported pain assessed after vaccination using a numerical rating scale (0-10)
Fear | immediately after vaccination (<5 minutes)
  self-reported fear assessed after vaccination using a numerical rating scale (0-10)

SECONDARY OUTCOMES:
Recruitment rate | before vaccination (1 day to 4 weeks)
  percentage of people eligible that participate
Feasibility of recruitment of subjects in the 2 study strata (i.e., preference to look or not look) | immediately before vaccination (<5 minutes)
  percentage of individuals that prefer to look or not look at baseline
Duration of appointment | immediately after vaccination
  Amount of time taken for appointment as per clock
Attrition of participants | immediately after vaccination
  number of participants that are lost/drop-out of study
Preferences of participants | immediately after vaccination (<5 minutes)
  participant preferences about interventions according to questionnaire
Fidelity of intervention | During vaccination
  Compliance with instruction to look at the needle or look away, according to checklist

CONTACTS AND LOCATIONS:
Locations (1):
- Anna Taddio, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mithal P, Simmons P, Cornelissen T, Wong H, Pillai Riddell R, McMurtry CM, Burry L, Stephens D, Taddio A. To look or not to look during vaccination: A pilot randomized trial. Can J Pain. 2018 Jan 5;2(1):1-8. doi: 10.1080/24740527.2017.1412254. eCollection 2018. PMID 35005359